CLINICAL TRIAL: NCT00151190
Title: Community Diabetes Education Program Evaluation
Brief Title: Community Diabetes Education Program Evaluation "Code Evaluation"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Institute for Faith Health Research of Dallas (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HSC-SPH-05-0092
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

INTERVENTIONS:
Behavioral: Education for diabetes self-management

SUMMARY:
The study is intended to determine the effectiveness and efficiency of a community diabetes education program administered by a community health worker in a low-cost community clinic. We expect an improvement in overall glycemic control in the experimental group of at least 20%. We also expect to document improvement in diabetes self-management skills, quality of life and an increase in achievement of ADA standards of care4 in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* people with no health insurance

Exclusion Criteria:

* people with any type of health insurance coverage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2005-04; Study Completion 2006-08

PRIMARY OUTCOMES:
HbA1c, Triglycerides, Cholesterol, Urine Microalbumin, Blood Pressure,

SECONDARY OUTCOMES:
Patients' attitudes and knowledge about diabetes self-management, American Diabetes Association standards of care.

CONTACTS AND LOCATIONS:
Overall Officials: DAN CULICA, MD, PhD, Principal Investigator — UTHSC School Public Health at Houston
Locations (1):
- Central Dallas Ministries Community Health Services Clinic, Dallas, Texas, United States

REFERENCES:
- [Derived] Prezio EA, Balasubramanian BA, Shuval K, Cheng D, Kendzor DE, Culica D. Evaluation of quality improvement performance in the Community Diabetes Education (CoDE) program for uninsured Mexican Americans: results of a randomized controlled trial. Am J Med Qual. 2014 Mar-Apr;29(2):124-34. doi: 10.1177/1062860613489165. Epub 2013 Jun 7. PMID 23748855
- [Derived] Prezio EA, Cheng D, Balasubramanian BA, Shuval K, Kendzor DE, Culica D. Community Diabetes Education (CoDE) for uninsured Mexican Americans: a randomized controlled trial of a culturally tailored diabetes education and management program led by a community health worker. Diabetes Res Clin Pract. 2013 Apr;100(1):19-28. doi: 10.1016/j.diabres.2013.01.027. Epub 2013 Feb 28. PMID 23453178